CLINICAL TRIAL: NCT02313909
Title: Multicenter, Randomized, Double-blind, Double-dummy, Active-comparator, Event-driven, Superiority Phase III Study of Secondary Prevention of Stroke and Prevention of Systemic Embolism in Patients With a Recent Embolic Stroke of Undetermined Source (ESUS), Comparing Rivaroxaban 15 mg Once Daily With Aspirin 100 mg
Brief Title: Rivaroxaban Versus Aspirin in Secondary Prevention of Stroke and Prevention of Systemic Embolism in Patients With Recent Embolic Stroke of Undetermined Source (ESUS)
Acronym: NAVIGATE ESUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted early due to no efficacy improvement over aspirin at an interim analysis and very little chance of showing overall benefit if study were completed
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry); Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16573; 2013-000768-27 (EudraCT Number)
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Stroke
Keywords: Rivaroxaban; Xarelto; Aspirin; Acetylsalicylic acid (ASA); Oral Anticoagulant; Blood Thinner; Stroke; Ischemic Stroke; Cryptogenic Stroke; Embolic stroke of undetermined source; ESUS; Transient Ischemic Attack; Thromboembolism; Cerebrovascular Disease
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemic Attack, Transient; Thromboembolism; Cerebrovascular Disorders | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban 15 mg orally once daily
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Other: Rivaroxaban-Placebo
- Aspirin (Active Comparator): Aspirin 100 mg orally once daily
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAY1019036); Other: Aspirin-Placebo

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15 mg, once daily, orally, tablet
  Arms: Rivaroxaban
Drug: Acetylsalicylic acid (Aspirin, BAY1019036) — 100 mg, once daily, orally, tablet
  Arms: Aspirin
Other: Rivaroxaban-Placebo — Matching placebo, once daily, orally, tablet
  Arms: Rivaroxaban
Other: Aspirin-Placebo — Matching placebo, once daily, orally, tablet
  Arms: Aspirin

SUMMARY:
This is a study in patients who recently had a brain attack (stroke) and in whom no clear cause of the stroke could be identified. These strokes are likely due to a blood clot and therefore, can be called embolic stroke of undetermined source. The abbreviation is ESUS. The study will compare 2 blood thinners. Patients will be randomly assigned to either Rivaroxaban 15 mg or Aspirin 100 mg and the study is intended to show, if patients given rivaroxaban have fewer blood clots in the brain (stroke) or in other blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Recent ESUS (between 7 days and 6 months), defined as:
* Recent ischemic stroke (including transient ischemic attack with positive neuroimaging) visualized by brain imaging that is not lacunar, and
* Absence of cervical carotid atherosclerotic stenosis> 50% or occlusion, and
* No atrial fibrillation after ≥ 24-hour cardiac rhythm monitoring, and
* No intra-cardiac thrombus on either transesophageal or transthoracic echocardiography, and
* No other specific cause of stroke (for example, arteritis, dissection, migraine/vasospasm, drug abuse)

Exclusion Criteria:

* Severely disabling stroke (modified Rankin score ≥4)
* Indication for chronic anticoagulation or antiplatelet therapy
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7213 (Actual)
Dates: Start 2014-12-23 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (374):
- United States (35):
  - Tucson, Arizona
  - Long Beach, California
  - Stanford, California
  - Torrance, California
  - New Haven, Connecticut
  - Gainesville, Florida
  - Joliet, Illinois
  - Iowa City, Iowa
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Mount Clemens, Michigan
  - New Brunswick, New Jersey
  - Buffalo, New York
  - New York, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Argentina (9):
  - Banfield, Buenos Aires
  - Ciudad Auton. de Buenos Aires, Buenos Aires
  - Mar del Plata, Buenos Aires
  - San Martín, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
  - Ciudad Auton. de Buenos Aires
  - Córdoba
  - Santa Fe
- Australia (10):
  - Camperdown, New South Wales
  - Waratah, New South Wales
  - Brisbane, Queensland
  - Southport, Queensland
  - Launceston, Tasmania
  - Clayton, Victoria
  - Footscray, Victoria
  - Murdoch, Western Australia
  - Elizabeth Vale
  - Nedlands
- Austria (9):
  - Klagenfurt, Carinthia
  - Villach, Carinthia
  - Bad Pirawarth, Lower Austria
  - Sankt Pölten, Lower Austria
  - Feldbach, Styria
  - Vöcklabruck, Upper Austria
  - Feldkirch, Vorarlberg
  - Salzburg
  - Vienna
- Belgium (7):
  - Bruges, West-Vlaanderen
  - Antwerp
  - Brussels
  - Bruxelles - Brussel
  - Dendermonde
  - Edegem
  - Hasselt
- Brazil (10):
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Joinville, Santa Catarina
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Matão, São Paulo
  - Ribeirão Preto, São Paulo
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (20):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Lethbridge, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Brandon, Manitoba
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Burlington, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
  - Québec
- Chile (7):
  - Los Ángeles, Bío-Bío
  - Osorno, Los Lagos Region
  - Port Montt, Los Lagos Region
  - Valdivia, Los Lagos Region
  - Viña del Mar, Región de Valparaíso
  - Santiago
  - Viña del Mar
- China (28):
  - Fuzhou, Fujian
  - Lanzhou, Gansu
  - Foshan, Guangdong
  - Guangzhou, Guangdong
  - Haikou, Hainan
  - Shijiazhuang, Hebei
  - Harbin, Heilongjiang
  - Zhengzhou, Henan
  - Wuhan, Hubei
  - Changsha, Hunan
  - Baotou, Inner Mongolia
  - Nantong, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shenyang, Liaoning
  - Qingdao, Shandong
  - Yantai, Shandong
  - Baoji, Shanxi
  - Xi’an, Shanxi
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
  - Taizhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Chongqing
  - Guangzhou
  - Shanghai
  - Tianjin
- Czechia (9):
  - Blansko
  - Brno
  - Hradec Králové
  - Jihlava
  - Olomouc
  - Ostrava Vitkovice
  - Ostrava-Poruba
  - Prague
  - Vyškov
- Denmark (6):
  - Aalborg
  - Aarhus C
  - Copenhagen
  - Glostrup Municipality
  - Herlev
  - Hillerød
- Finland (7):
  - Helsinki
  - Lappeenranta
  - OYS
  - Sairaalamäki
  - Tampere
  - Turku
  - Vaasa
- France (12):
  - Antony
  - Bordeaux
  - Brest
  - Caen
  - Dijon
  - Le Chesnay
  - Limoges
  - Nantes
  - Nîmes
  - Paris
  - Saint-Priest-en-Jarez
  - Strasbourg
- Germany (16):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Würzburg, Bavaria
  - Hanover, Lower Saxony
  - Düsseldorf, North Rhine-Westphalia
  - Meerbusch, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Dresden, Saxony
  - Markkleeberg, Saxony
  - Wermsdorf, Saxony
  - Halle, Saxony-Anhalt
  - Altenburg, Thuringia
  - Berlin
  - Hamburg
- Greece (4):
  - Athens
  - Ioannina
  - Larissa
  - Thessaloniki
- Hungary (11):
  - Budapest
  - Debrecen
  - Eger
  - Győr
  - Kistarcsa
  - Miskolc
  - Nagykanizsa
  - Nyíregyháza
  - Sopron
  - Szeged
  - Zalaegerszeg
- Ireland (2):
  - Dublin
  - Galway
- Israel (7):
  - Ashkelon
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (12):
  - L’Aquila, Abruzzo
  - Vibo Valentia, Calabria
  - Parma, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Rome, Lazio
  - Milan, Lombardy
  - Pavia, Lombardy
  - Isernia, Molise
  - Cagliari, Sardinia
  - Ancona, The Marches
  - Perugia, Umbria
  - Verona, Veneto
- Japan (35):
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Seto, Aichi-ken
  - Toyota, Aichi-ken
  - Kitakyushu, Fukuoka
  - Kōriyama, Fukushima
  - Fukuyama, Hiroshima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Kushiro, Hokkaido
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Isehara, Kanagawa
  - Kawasaki, Kanagawa
  - Sendai, Miyagi
  - Sasebo, Nagasaki
  - Tenri, Nara
  - Kurashiki, Okayama-ken
  - Matsubara, Osaka
  - Sakai, Osaka
  - Suita, Osaka
  - Hidaka, Saitama
  - Bunkyo-ku, Tokyo
  - Hachiōji, Tokyo
  - Kodaira, Tokyo
  - Musashino, Tokyo
  - Shinjuku-ku, Tokyo
  - Sumida-ku, Tokyo
  - Fukuoka
  - Hiroshima
  - Kakogawa
  - Kochi
  - Kyoto
  - Niigata
  - Okayama
- Mexico (8):
  - Gustavo Adolfo Madero, Mexico City
  - México, D.F., Mexico City
  - Morelia, Michoacán
  - México D.F., México
  - Monterrey, Nuevo León
  - Mérida, Yucatán
  - Aguascalientes
  - México D.F.
- Poland (11):
  - Bialystok
  - Chełm
  - Gdansk
  - Gmina Końskie
  - Katowice
  - Lodz
  - Olsztyn
  - Sandomierz
  - Siedlce
  - Skarżysko-Kamienna
  - Warsaw
- Portugal (7):
  - Vilanova de Gaia, Porto District
  - Almada
  - Amadora
  - Coimbra
  - Lisbon
  - Porto
  - Vila Franca de Xira
- Russia (12):
  - Chelyabinsk
  - Kaluga
  - Kazan'
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Tomsk
  - Ulyanovsk
  - Volgograd
  - Yaroslavl
  - Yekaterinburg
- South Africa (3):
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Durban
- South Korea (9):
  - Donggu, Gwangju Gwang''yeogsi
  - Anyang-si, Gyeonggido
  - Goyang, Gyeonggido
  - Seongnam-si, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daegu
  - Incheon
  - Seoul
- Spain (20):
  - Santiago de Compostela, A Coruña
  - Badalona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Sant Joan Despí, Barcelona
  - Castellon, Castellón
  - El Palmar (Murcia), Murcia
  - A Coruña
  - Badajoz
  - Barcelona
  - Bilbao
  - Cáceres
  - Girona
  - Granada
  - León
  - Lleida
  - Madrid
  - Seville
  - Valencia
  - Valladolid
  - Zaragoza
- Sweden (5):
  - Gothenburg
  - Hässleholm
  - Lund
  - Malmo
  - Umeå
- Switzerland (8):
  - Aarau, Canton of Aargau
  - Basel, Canton of Basel-City
  - Lugano, Canton Ticino
  - Baden
  - Bern
  - Fribourg
  - Geneva
  - Zurich
- Turkey (Türkiye) (5):
  - Ankara
  - Antakya
  - Istanbul
  - Kahramanmaraş
  - Konya
- United Kingdom (30):
  - High Wycombe, Buckinghamshire
  - Milton Keynes, Buckinghamshire
  - Cambridge, Cambridgeshire
  - Exeter, Devon
  - Colchester, Essex
  - Westcliff-on-Sea, Essex
  - Gloucester, Gloucestershire
  - Watford, Hertfordshire
  - Ashford, Kent
  - Margate, Kent
  - Leicester, Leicestershire
  - Boston, Lincolnshire
  - Harrow, London
  - Great Yarmouth, Norfolk
  - Taunton, Somerset
  - Yeovil, Somerset
  - Sheffield, South Yorkshire
  - Stoke-on-Trent, Staffordshire
  - Glasgow, Stratchclyde
  - Gateshead, Tyne and Wear
  - Sunderland, Tyne and Wear
  - Wolverhampton, West Midlands
  - Leeds, West Yorkshire
  - Salisbury, Wiltshire
  - Aberdeen
  - Durham
  - Edinburgh
  - London
  - Luton
  - Norwich

REFERENCES:
- [Result] Hart RG, Sharma M, Mundl H, Kasner SE, Bangdiwala SI, Berkowitz SD, Swaminathan B, Lavados P, Wang Y, Wang Y, Davalos A, Shamalov N, Mikulik R, Cunha L, Lindgren A, Arauz A, Lang W, Czlonkowska A, Eckstein J, Gagliardi RJ, Amarenco P, Ameriso SF, Tatlisumak T, Veltkamp R, Hankey GJ, Toni D, Bereczki D, Uchiyama S, Ntaios G, Yoon BW, Brouns R, Endres M, Muir KW, Bornstein N, Ozturk S, O'Donnell MJ, De Vries Basson MM, Pare G, Pater C, Kirsch B, Sheridan P, Peters G, Weitz JI, Peacock WF, Shoamanesh A, Benavente OR, Joyner C, Themeles E, Connolly SJ; NAVIGATE ESUS Investigators. Rivaroxaban for Stroke Prevention after Embolic Stroke of Undetermined Source. N Engl J Med. 2018 Jun 7;378(23):2191-2201. doi: 10.1056/NEJMoa1802686. Epub 2018 May 16. PMID 29766772
- [Result] Kasner SE, Lavados P, Sharma M, Wang Y, Wang Y, Davalos A, Shamalov N, Cunha L, Lindgren A, Mikulik R, Arauz A, Lang W, Czlonkowska A, Eckstein J, Gagliardi R, Amarenco P, Ameriso SF, Tatlisumak T, Veltkamp R, Hankey GJ, Toni DS, Bereczki D, Uchiyama S, Ntaios G, Yoon BW, Brouns R, DeVries Basson MM, Endres M, Muir K, Bornstein N, Ozturk S, O'Donnell M, Mundl H, Pater C, Weitz J, Peacock WF, Swaminathan B, Kirsch B, Berkowitz SD, Peters G, Pare G, Themeles E, Shoamanesh A, Connolly SJ, Hart RG; NAVIGATE ESUS Steering Committee and Investigators. Characterization of Patients with Embolic Strokes of Undetermined Source in the NAVIGATE ESUS Randomized Trial. J Stroke Cerebrovasc Dis. 2018 Jun;27(6):1673-1682. doi: 10.1016/j.jstrokecerebrovasdis.2018.01.027. Epub 2018 Mar 7. PMID 29525076
- [Result] Hart RG, Sharma M, Mundl H, Shoamanesh A, Kasner SE, Berkowitz SD, Pare G, Kirsch B, Pogue J, Pater C, Peters G, Davalos A, Lang W, Wang Y, Wang Y, Cunha L, Eckstein J, Tatlisumak T, Shamalov N, Mikulik R, Lavados P, Hankey GJ, Czlonkowska A, Toni D, Ameriso SF, Gagliardi RJ, Amarenco P, Bereczki D, Uchiyama S, Lindgren A, Endres M, Brouns R, Yoon BW, Ntaios G, Veltkamp R, Muir KW, Ozturk S, Arauz A, Bornstein N, Bryer A, O'Donnell MJ, Weitz J, Peacock F, Themeles E, Connolly SJ. Rivaroxaban for secondary stroke prevention in patients with embolic strokes of undetermined source: Design of the NAVIGATE ESUS randomized trial. Eur Stroke J. 2016 Sep;1(3):146-154. doi: 10.1177/2396987316663049. Epub 2016 Aug 3. PMID 31008276
- [Derived] Lee SF, Whiteley W, Bosch J, Sherlock L, Cukierman-Yaffe T, O'Donnell M, Eikelboom JW, Gerstein HC, Bangdiwala SI, Muniz-Terrera G. Improving analysis of cognitive outcomes in cardiovascular trials using different statistical approaches. Trials. 2024 Oct 2;25(1):644. doi: 10.1186/s13063-024-08482-2. PMID 39358761
- [Derived] Sharma M, Smith EE, Pearce LA, Perera KS, Kasner SE, Yoon BW, Ameriso SF, Puig J, Damgaard D, Fiebach JB, Muir KW, Veltkamp RC, Toni DS, Shamalov N, Gagliardi RJ, Mikulik R, Engelter ST, Bereczki D, O'Donnell MJ, Saad F, Shoamanesh A, Berkowitz SD, Mundl H, Hart RG; NAVIGATE ESUS MRI Substudy Investigators. Rivaroxaban versus aspirin for prevention of covert brain infarcts in patients with embolic stroke of undetermined source: NAVIGATE ESUS MRI substudy. Int J Stroke. 2022 Aug;17(7):799-805. doi: 10.1177/17474930211058012. Epub 2021 Nov 18. PMID 34791941
- [Derived] Merkler AE, Pearce LA, Kasner SE, Shoamanesh A, Birnbaum LA, Kamel H, Sheth KN, Sharma R. Left Ventricular Dysfunction Among Patients With Embolic Stroke of Undetermined Source and the Effect of Rivaroxaban vs Aspirin: A Subgroup Analysis of the NAVIGATE ESUS Randomized Clinical Trial. JAMA Neurol. 2021 Dec 1;78(12):1454-1460. doi: 10.1001/jamaneurol.2021.3828. PMID 34694346
- [Derived] Sharma M, Smith EE, Pearce LA, Shoamanesh A, Perera KS, Coutts SB, Damgaard D, Ameriso SF, Rha JH, Modrau B, Yoon BW, Romano M, Messe SR, Barlinn J, Lambeck J, Saad F, Berkowitz SD, Mundl H, Connolly SJ, Hart RG; NAVIGATE ESUS MIND MRI Substudy Investigators. Frequency and Patterns of Brain Infarction in Patients With Embolic Stroke of Undetermined Source: NAVIGATE ESUS Trial. Stroke. 2022 Jan;53(1):45-52. doi: 10.1161/STROKEAHA.120.032976. Epub 2021 Sep 20. PMID 34538089
- [Derived] Shoamanesh A, Hart RG, Connolly SJ, Kasner SE, Smith EE, Marti-Fabregas J, Liu YY, Uchiyama S, Mikulik R, Veltkamp R, O'Donnell MJ, Ntaios G, Muir KW, Field TS, Santo GC, Olavarria V, Mundl H, Lutsep H, Berkowitz SD, Sharma M. Microbleeds and the Effect of Anticoagulation in Patients With Embolic Stroke of Undetermined Source: An Exploratory Analysis of the NAVIGATE ESUS Randomized Clinical Trial. JAMA Neurol. 2021 Jan 1;78(1):11-20. doi: 10.1001/jamaneurol.2020.3836. PMID 33074284
- [Derived] Scheitz JF, Pare G, Pearce LA, Mundl H, Peacock WF, Czlonkowska A, Sharma M, Nolte CH, Shoamanesh A, Berkowitz SD, Krahn T, Endres M; NAVIGATE-ESUS Biomarker Working Group. High-Sensitivity Cardiac Troponin T for Risk Stratification in Patients With Embolic Stroke of Undetermined Source. Stroke. 2020 Aug;51(8):2386-2394. doi: 10.1161/STROKEAHA.120.029628. Epub 2020 Jul 9. PMID 32640945
- [Derived] Veltkamp R, Pearce LA, Korompoki E, Sharma M, Kasner SE, Toni D, Ameriso SF, Mundl H, Tatlisumak T, Hankey GJ, Lindgren A, Berkowitz SD, Arauz A, Ozturk S, Muir KW, Chamorro A, Perera K, Shuaib A, Rudilosso S, Shoamanesh A, Connolly SJ, Hart RG. Characteristics of Recurrent Ischemic Stroke After Embolic Stroke of Undetermined Source: Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2020 Oct 1;77(10):1233-1240. doi: 10.1001/jamaneurol.2020.1995. PMID 32628266
- [Derived] Mikulik R, Eckstein J, Pearce LA, Mundl H, Rudilosso S, Olavarria VV, Shoamanesh A, Chamorro A, Marti-Fabregas J, Veltkamp R, Ozturk S, Tatlisumak T, Peacock WF, Berkowitz SD, Connolly SJ, Hart RG. Frequency and Predictors of Major Bleeding in Patients With Embolic Strokes of Undetermined Source: NAVIGATE-ESUS Trial. Stroke. 2020 Jul;51(7):2139-2147. doi: 10.1161/STROKEAHA.119.027995. Epub 2020 Jun 10. PMID 32517582
- [Derived] Ntaios G, Pearce LA, Veltkamp R, Sharma M, Kasner SE, Korompoki E, Milionis H, Mundl H, Berkowitz SD, Connolly SJ, Hart RG; NAVIGATE ESUS Investigators. Potential Embolic Sources and Outcomes in Embolic Stroke of Undetermined Source in the NAVIGATE-ESUS Trial. Stroke. 2020 Jun;51(6):1797-1804. doi: 10.1161/STROKEAHA.119.028669. Epub 2020 Apr 16. PMID 32295509
- [Derived] Martinez-Majander N, Ntaios G, Liu YY, Ylikotila P, Joensuu H, Saarinen J, Perera KS, Marti-Fabregas J, Chamorro A, Rudilosso S, Prats-Sanchez L, Berkowitz SD, Mundl H, Themeles E, Tiainen M, Demchuk A, Kasner SE, Hart RG, Tatlisumak T; NAVIGATE ESUS investigators. Rivaroxaban versus aspirin for secondary prevention of ischaemic stroke in patients with cancer: a subgroup analysis of the NAVIGATE ESUS randomized trial. Eur J Neurol. 2020 May;27(5):841-848. doi: 10.1111/ene.14172. Epub 2020 Mar 11. PMID 32056346
- [Derived] Ntaios G, Pearce LA, Meseguer E, Endres M, Amarenco P, Ozturk S, Lang W, Bornstein NM, Molina CA, Pagola J, Mundl H, Berkowitz SD, Liu YY, Sen S, Connolly SJ, Hart RG. Aortic Arch Atherosclerosis in Patients With Embolic Stroke of Undetermined Source: An Exploratory Analysis of the NAVIGATE ESUS Trial. Stroke. 2019 Nov;50(11):3184-3190. doi: 10.1161/STROKEAHA.119.025813. Epub 2019 Sep 17. PMID 31526123
- [Derived] Ntaios G, Swaminathan B, Berkowitz SD, Gagliardi RJ, Lang W, Siegler JE, Lavados P, Mundl H, Bornstein N, Meseguer E, Amarenco P, Cucchiara B, Camps-Renom P, Makaritsis K, Korompoki E, Papavasileiou V, Marti-Fabregas J, Milionis H, Vemmos K, Connolly SJ, Hart RG; NAVIGATE ESUS Investigators. Efficacy and Safety of Rivaroxaban Versus Aspirin in Embolic Stroke of Undetermined Source and Carotid Atherosclerosis. Stroke. 2019 Sep;50(9):2477-2485. doi: 10.1161/STROKEAHA.119.025168. Epub 2019 Aug 12. PMID 31401971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 31 countries between 23 December 2014 (first participant first visit) and 15 February 2018 (last participant last visit).
Pre-assignment Details: Overall, 7582 participants were screened; of these 369 participants were screen failures. A total of 7213 participants were randomized, of which 92 never took study drug; 3562 were treated with rivaroxaban(Xarelto, BAY59-7939) /placebo and 3559 were treated with acetylsalicylic acid/placebo.
Groups:
- Rivaroxaban 15 mg OD: Subjects received rivaroxaban 15 mg immediate-release film-coated tablet and matching placebo of acetylsalicylic acid orally once daily (OD).
- Acetylsalicylic Acid 100 mg OD: Subjects received acetylsalicylic acid 100 mg enteric-coated tablet and matching placebo of rivaroxaban orally once daily (OD).
Period: Overall Study
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Started | 3609 | 3604
Treated | 3562 | 3559
Completed | 3552 | 3554
Not Completed | 57 | 50
Not completed — Consent withdrawn by participant | 33 | 33
Not completed — Lost to Follow-up | 24 | 17

BASELINE CHARACTERISTICS:
Population: Intention-to-treat analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD | Total
Number analyzed (Participants) | 3609 | 3604 | 7213
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.8) | 66.9 (9.8) | 66.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1377 | 1400 | 2777
  Male | 2232 | 2204 | 4436
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intention-to-treat analysis set included all randomized participants.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 716 | 698 | 1414
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 51 | 60 | 111
    White | 2613 | 2605 | 5218
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 229 | 241 | 470
Stroke or TIA (prior to qualifying stroke) or Other medical history [Number; unit: count of participants] — TIA: Transient Ischemic Attack
  count of participants
    Stroke or TIA | 620 | 643 | 1263
    Other medical history | 2989 | 2961 | 5950
Time from qualifying stroke to randomization [Median (Inter-Quartile Range); unit: days] — Population: Intention-to-treat analysis set included all randomized participants.
  days | 38.0 [15.0 to 89.0] | 36.0 [14.0 to 86.5] | 37.0 [14.0 to 88.0]

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of the Composite Efficacy Outcome (Adjudicated)
Description: Components of composite efficacy outcome (adjudicated) includes stroke (ischemic, hemorrhagic, and undefined stroke, TIA with positive neuroimaging) and systemic embolism. Incidence rate estimated as number of participants with incident events divided by cumulative at-risk time, where participant is no longer at risk once an incident event occurred.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: Intention-to-treat analysis set included all randomized participants. Participants who were evaluable for this measure at given time period for the arm were included in the category.
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 5.14 [4.40 to 5.97] | 4.78 [4.07 to 5.58]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis: Stroke + Systemic embolism: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.51884, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.87 to 1.33]

2. Primary Outcome: Incidence Rate of a Major Bleeding Event According to the International Society on Thrombosis and Haemostasis (ISTH) Criteria (Adjudicated)
Description: Major bleeding event (as per ISTH), defined as bleeding event that met at least one of following: fatal bleeding; symptomatic bleeding in a critical area or organ (intraarticular, intramuscular with compartment syndrome, intraocular, intraspinal, pericardial, or retroperitoneal); symptomatic intracranial haemorrhage; clinically overt bleeding associated with a recent decrease in the hemoglobin level of greater than or equal to (>=) 2 grams per decilitre (g/dL) (20 grams per liter [g/L]; 1.24 millimoles per liter [mmol/L]) compared to the most recent hemoglobin value available before the event; clinically overt bleeding leading to transfusion of 2 or more units of packed red blood cells or whole blood. The results were based on classification of events that have been positively adjudicated as major bleeding events. Incidence rate estimated as number of subjects with incident events divided by cumulative at-risk time, where subject is no longer at risk once an incident event occurred.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 1.82 [1.39 to 2.33] | 0.67 [0.42 to 1.00]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis: ISTH major bleeding events: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.00002, Log Rank; Hazard Ratio (HR) = 2.72, 95% CI 2-sided [1.68 to 4.39]

3. Secondary Outcome: Incidence Rate of Any of the Following: Cardiovascular Death, Recurrent Stroke, Systemic Embolism and Myocardial Infarction
Description: Incidence rate estimated as number of participants with incident events divided by cumulative at-risk time, where participant is no longer at risk once an incident event occurred. Cardiovascular death includes death due to hemorrhage and death with undetermined/unknown cause. Systemic embolism is defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms. The diagnosis of myocardial infarction requires the combination of: 1)evidence of myocardial necrosis (either changes in cardiac biomarkers or post-mortem pathological findings); and 2)supporting information derived from the clinical presentation, electrocardiographic changes, or the results of myocardial or coronary artery imaging.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 6.20 [5.38 to 7.10] | 5.85 [5.05 to 6.73]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Confidence intervals were calculated, if at least 1 event in each treatment arm existed. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.56922, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.87 to 1.29]

4. Secondary Outcome: Incidence Rate of All-Cause Mortality
Description: All-cause mortality includes all deaths of participants due to any cause.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 1.88 [1.45 to 2.40] | 1.50 [1.12 to 1.97]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Confidence intervals were calculated, if at least 1 event in each treatment arm existed. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.22078, Log Rank; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.87 to 1.81]

5. Secondary Outcome: Incidence Rate of the Following: Stroke, Ischemic Stroke, Disabling Stroke, Cardiovascular (CV) Death, Myocardial Infarction
Description: Disabling stroke is defined as stroke with modified Rankin score (mRS) greater than or equal to (>=) 4 as assessed by investigator. mRS spans 0-6, running from perfect health to death. A score of 0-3 indicates functional status ranging from no symptoms to "moderate disability" (defined in the mRS as requiring some help, but able to walk without assistance); mRS 4-6 indicates functional status ranging from "moderately severe disability" (unable to walk or to attend to own bodily needs without assistance)through to death. CV death includes death due to hemorrhage and death with undetermined/unknown cause. Diagnosis of myocardial infarction requires combination of: 1) evidence of myocardial necrosis either changes in cardiac biomarkers or post-mortem pathological findings); 2) supporting information derived from clinical presentation, electrocardiographic changes, or results of myocardial or coronary artery imaging.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years
  Stroke | 5.11 [4.37 to 5.93] | 4.71 [4.01 to 5.51]
  Ischemic stroke | 4.71 [4.01 to 5.51] | 4.56 [3.87 to 5.34]
  Disabling stroke | 1.20 [0.86 to 1.62] | 0.84 [0.56 to 1.21]
  CV death(includes death due to hemorrhage) | 0.99 [0.68 to 1.38] | 0.66 [0.42 to 1.00]
  Myocardial infarction | 0.49 [0.29 to 0.79] | 0.67 [0.42 to 1.00]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis 1: Stroke: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.47970, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.87 to 1.34]
Statistical Analysis 2: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis 2: Ischemic stroke: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.78738, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.83 to 1.29]
Statistical Analysis 3: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis 3: Disabling stroke: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.14822, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.88 to 2.28]
Statistical Analysis 4: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis 4:CV death: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.14051, Log Rank; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [0.87 to 2.52]
Statistical Analysis 5: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis 5: Myocardial infarction: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.34284, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.39 to 1.38]

6. Secondary Outcome: Incidence Rate of Life-Threatening Bleeding Events
Description: Life-threatening bleeding was defined as a subset of major bleeding that met at least one of the following criteria: 1) fatal bleeding; 2) symptomatic intracranial haemorrhage; 3) reduction in hemoglobin of at least 5 g/dl (50 g/l; 3.10 mmol/L); 4) transfusion of at least 4 units of packed red cells or whole blood; 5) associated with hypotension requiring the use of intravenous inotropic agents; 6) necessitated surgical intervention. Incidence rate estimated as number of participants with incident events divided by cumulative at-risk time, where participant is no longer at risk once an incident event occurred.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 1.02 [0.71 to 1.42] | 0.43 [0.24 to 0.72]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.00443, Log Rank; Hazard Ratio (HR) = 2.34, 95% CI 2-sided [1.28 to 4.29]

7. Secondary Outcome: Incidence Rate of Clinically Relevant Non-Major Bleeding Events
Description: Non-major clinically relevant bleeding was defined as non-major overt bleeding but required medical attention (example: hospitalization, medical treatment for bleeding), and/or was associated with the study drug interruption of more than 14 days. The results were based on the outcome events at or after randomization until the efficacy cut-off date. Incidence rate estimated as number of participants with incident events divided by cumulative at-risk time, where participant is no longer at risk once an incident event occurred.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 3.52 [2.91 to 4.21] | 2.32 [1.84 to 2.90]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.00451, Log Rank; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [1.13 to 2.00]

8. Secondary Outcome: Incidence Rate of Intracranial Hemorrhage
Description: Intracranial hemorrhage included all bleeding events that occurred in intracerebral, sub arachnoidal as well as subdural or epidural sites. The below table displays results for all randomized participants and the outcomes at or after randomization until the efficacy cut-off date. Incidence rate estimated as number of participants with incident events divided by cumulative at-risk time, where participant is no longer at risk once an incident event occurred.
Time Frame: From randomization until the efficacy cut-off date (median 326 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event/100 participant-years
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
Number analyzed (Participants) | 3609 | 3604
event/100 participant-years | 0.70 [0.45 to 1.04] | 0.35 [0.18 to 0.61]
Statistical Analysis 1: Comparison: Rivaroxaban 15 mg OD vs Acetylsalicylic Acid 100 mg OD; Statistical analysis 1: Risk reduction was estimated with the stratified Cox proportional hazards model. Hazard ratios (95% confidence interval) as compared to acetylsalicylic acid arm were reported. Rivaroxaban treatment was compared with the Acetylsalicylic acid control group using a stratified log-rank test. P-values (two-sided) as compared to acetylsalicylic acid arm were based on the log-rank test; Test type: Superiority; p = 0.04409, Log Rank; Hazard Ratio (HR) = 2.01, 95% CI 2-sided [1.00 to 4.02]

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 2 days after the last dose of study drug, an average of 279 days
Description: Safety analysis set included all randomized participants who received at least one dose of study drug.
Arm/Group | Rivaroxaban 15 mg OD | Acetylsalicylic Acid 100 mg OD
All-Cause Mortality (participants affected / at risk) | 73/3562 | 58/3559
Serious Adverse Events (participants affected / at risk) | 466/3562 | 434/3559
Other Adverse Events (participants affected / at risk) | 308/3562 | 294/3559
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 15 mg OD (N=3562) | Acetylsalicylic Acid 100 mg OD (N=3559)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 3 (3)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 36 (36) | 37 (37)
Atrial flutter (Cardiac disorders) | 5 (5) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac amyloidosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 3 (3)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 3 (3)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Endocarditis noninfective (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pulmonary arteriovenous fistula (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 4 (5) | 8 (10)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Ophthalmic vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 7 (7) | 5 (5)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastric volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 4 (4) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 6 (6) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Corneal graft rejection (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Corneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 6 (6) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 2 (2) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14) | 14 (14)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 6 (7)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 4 (5)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 (4) | 0 (0)
Neurocysticercosis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (2) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Incorrect dosage administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 6 (6)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (12) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colorectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 8 (8)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Chorea (Nervous system disorders) | 1 (1) | 0 (0)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 7 (8) | 8 (8)
Facial paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Hemiparesis (Nervous system disorders) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 4 (4)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 9 (10) | 9 (9)
Status epilepticus (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 10 (10) | 8 (8)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 2 (2)
Partial seizures (Nervous system disorders) | 5 (5) | 2 (2)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Central pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke seizure (Nervous system disorders) | 0 (0) | 2 (3)
Hemianaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pseudostroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparaesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 1 (1)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Completed suicide (Psychiatric disorders) | 0 (0) | 2 (2)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive-compulsive personality disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic reaction (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Neurologic somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Costovertebral angle tenderness (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 6 (6)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Atrial septal defect repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 3 (3) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 6 (6)
Hypertensive crisis (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 5 (5) | 5 (6)
May-Thurner syndrome (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 15 mg OD (N=3562) | Acetylsalicylic Acid 100 mg OD (N=3559)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 60 (60) | 60 (60)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Fabry's disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 7 (7)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (4)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 4 (4)
Chills (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 1 (3)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inappropriate schedule of drug administration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 10 (10) | 9 (9)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Labelled drug-drug interaction medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dosage administered (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Medication monitoring error (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Intentional product misuse (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Coagulation factor VIII level increased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Visual acuity tests abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Haemochromatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6) | 7 (7)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 10 (10) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 3 (4)
Vertebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hyposmia (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Impatience (Psychiatric disorders) | 1 (1) | 0 (0)
Abulia (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Post stroke depression (Psychiatric disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 2 (2) | 5 (5)
Tooth extraction (Surgical and medical procedures) | 2 (3) | 2 (2)
Cataract operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Implantable cardiac monitor insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 11 (11) | 7 (8)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 2 (2)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to no efficacy improvement over aspirin at the second interim analysis and very little chance of showing overall benefit if the study were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Global PI to provide to Bayer for review any proposed Publication/oral presentation relating to Study/Study Drug/Results at least 20 days prior to submission or presentation of the Publication. Abstracts/posters/oral presentations to be provided to Bayer 5 working days before Publication/presentation. Bayer may provide comments within the applicable period. Under certain circumstances Bayer may request a further delay of publications to avoid adverse effects on a Bayer patent application.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT02313909/SAP_000.pdf
  • Study Protocol (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT02313909/Prot_001.pdf